CLINICAL TRIAL: NCT06519786
Title: Safety and Efficacy of Metformin for Treatment of Cytopenia in Children and Adolescents With Fanconi Anemia
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: FMASU MD 274/2022
Record Dates: First submitted 2023-12-27; First posted 2024-07-25 (Actual); Last update posted 2024-07-25 (Actual); Status verified 2023-12

CONDITIONS: Fanconi Anemia
MeSH Terms: conditions — Fanconi Anemia | interventions — Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Metformin group (Experimental): Patients will receive metformin immediate-release tablets orally for 24 weeks. Starting dose will be 500 mg once daily for all patients and the dose will be increased by 500 mg weekly until the goal dose is achieved (500 mg twice daily for patients < 10 years of age, and 1000 mg twice daily for patients 10 years or older).
  Interventions: Drug: Metformin
- Other treatment group (No Intervention): Patients will receive supportive treatment as indicated

INTERVENTIONS:
Drug: Metformin — Patients will receive metformin immediate-release tablets orally for 24 weeks. Starting dose will be 500 mg once daily for all patients and the dose will be increased by 500 mg weekly until the goal dose is achieved (500 mg twice daily for patients < 10 years of age, and 1000 mg twice daily for patients 10 years or older)
  Other Names: Glucophage
  Arms: Metformin group

SUMMARY:
Prospective interventional open-label non-randomized controlled trial to assess safety and efficacy of metformin in treating cytopenia in children and adolescents with Fanconi Anemia.

DETAILED DESCRIPTION:
Fanconi anemia (FA) is a genetic disease characterized by bone marrow failure, cancer susceptibility, and developmental abnormalities. Allogeneic hematopoietic stem cell transplantation offers curative therapy for hematologic complications of FA.

Oxymetholone is commonly used in the management of FA as it improves blood counts, red cells, and platelets. However, its use is limited by its high toxicity profile.

Metformin is a potential agent that reduces levels of both chromosomal radials and breaks in FA cells and increases the size of the hematopoietic stem cell compartment thus reducing cytopenia in patients with FA.

ELIGIBILITY:
Inclusion Criteria:

* Age: 5 to 18 years
* Patients who are diagnosed with Fanconi anemia based on clinical features and confirmed by increased chromosomal breakage on diepoxybutane (DEB) stress testing.
* Presence of cytopenia (at least one of the following: hemoglobin (Hb) < 10 g/dL, platelet count < 100 x 109/L, or an absolute neutrophil count (ANC) < 1.0 x 109/L
* Patients receiving other therapies e.g., androgens are eligible for enrollment after a one-month washout period before the start of metformin.

Exclusion Criteria:

* Patients who underwent bone marrow transplantation.
* Patients with evidence of myelodysplasia, leukemia, or other concurrent malignancy.
* Patients who have a history of allergic reactions to metformin or similar compounds.
* Patients with a history of symptomatic hypoglycemia over the past year or hypoglycemia < 50 mg/dL on screening and baseline laboratory assessments.
* Patients with type 1 diabetes mellitus.
* Patients with vitamin B12 deficiency.
* Patients with Glucose-6-Phosphate Dehydrogenase deficiency.
* Patients with abnormal Kidney function tests including serum creatinine, elevated liver function tests including live enzymes (ALT or AST > 135 U/L, total bilirubin > 1.5 x upper limit of normal for age, and/or patients with metabolic acidosis (bicarbonate < 17 meq/L on venous blood gases).

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-10-05 (Actual); Primary Completion 2024-10 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Hematologic response (erythroid) | 24 weeks
  Erythroid response (pretreatment, < 11 g/dL): Hgb increase by > 1.5 g/dL or Relevant reduction of units of RBC transfusions by an absolute number of at least 4 RBC transfusions/8 wk compared with the pretreatment transfusion number in the previous 8 wk.
Hematologic response (platelets) | 24 weeks
  Platelet response (pretreatment, < 100x10e9/L): Absolute increase of > 30 x 10e9/L for patients starting with > 20 x 10e9/L platelets or Increase from < 20 x 10e9/L to > 20 x10e9/L and by at least 100%
Hematologic response (Neutrophil count) | 24 weeks
  Neutrophil response (pretreatment, < 1.0 x 10e9/L): At least 100% increase and an absolute increase > 0.5 x 10e9/L

CONTACTS AND LOCATIONS:
Locations (2):
- Egypt (2):
  - University of Alexandria, Alexandria
  - Ain Shams University, Cairo